CLINICAL TRIAL: NCT04754815
Title: Phase II Study of Pemetrexed or Nab-paclitaxel With Pembrolizumab in Elderly (>/= 75 Years) Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of Pembrolizumab With Single Agent Chemotherapy in Elderly Patients With Advanced NSCLC
Acronym: HFHS 21-01
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Logistical challenges primarily due to COVID led to delay in starting the study and now is not felt to be clinically relevant.
Sponsor: Shirish Gadgeel (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Shirish Gadgeel, Principle Investigator, Henry Ford Health System
Organization: Henry Ford Health System (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFHS 21-01
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2021-02

CONDITIONS: Non Small Cell Lung Cancer; Advanced Lung Non-Small Cell Carcinoma; PD-L1 Gene Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Pemetrexed; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: Single arm open label with 2 treatment options
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pembrolizumab + Pemetrexed (Experimental): Pembrolizumab 200mg intravenous (IV) infusion on Day 1 of each 21 day cycle. Treatment repeats every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity + pemetrexed 500mg intravenous (IV) infusion (with vitamin supplementation) on Day 1 of each 21 day cycle up to 35 cycles or until disease progression.
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed; Other: Laboratory Biomarker Analysis
- Pembrolizumab + Paclitaxel OR Paclitaxel (Experimental): Pembrolizumab 200mg intravenous (IV) infusion on Day 1 of each 21 day cycle. Treatment repeats every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity
  + Paclitaxel 100 mg/m2 intravenous (IV) infusion on days 1 and 8 of each 21 day treatment cycle
  OR Paclitaxel100 mg/m2 intravenous (IV) infusion on days 1 and 8 of each 21 day treatment cycle until disease progression.
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel; Drug: Nab-paclitaxel; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Pembrolizumab — PD-L1 inhibitor administered as an intravenous (IV) infusion.
  Other Names: Keytruda
Drug: Pemetrexed — Folate analog metabolic inhibitor administered as an intravenous (IV) infusion single agent chemotherapy for advanced NSCLC
  Other Names: ALIMTA
  Arms: Pembrolizumab + Pemetrexed
Drug: Paclitaxel — A novel antimicrotubular agent administered as an intravenous (IV) infusion single agent chemotherapy for advanced NSCLC
  Other Names: TAXOL
  Arms: Pembrolizumab + Paclitaxel OR Paclitaxel
Drug: Nab-paclitaxel — Microtubule inhibitor administered as an intravenous (IV) infusion indicated for the treatment of locally advanced or metastatic NSCLC
  Other Names: ABRAXANE®
  Arms: Pembrolizumab + Paclitaxel OR Paclitaxel
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This Phase II trial is to see how well single agent chemotherapy and pembrolizumab work elderly patients (≥ 75 years) with advanced non small cell lung cancer (NSCLC). Pembrolizumab stimulates your immune system to help fight lung cancer. This treatment approach may be better tolerated in elderly patients.

DETAILED DESCRIPTION:
Primary Objective(s), Hypothesis(es), and Endpoint(s)

I. Objective: To evaluate the efficacy of single agent chemotherapy and pembrolizumab in elderly (≥ 75 years) advanced NSCLC patients Hypothesis: We propose that single agent chemotherapy with pembrolizumab will be better tolerated and will provide similar efficacy as platinum-based combination chemotherapy with pembrolizumab in advanced elderly (≥75 years) NSCLC patients.

Primary Endpoint:

I. Assess median PFS in elderly (≥ 75 years) advanced NSCLC patients with tumor PD-L1 (<50%) treated with pemetrexed or nab-paclitaxel and pembrolizumab.

Secondary Objective(s), Hypothesis(es), and Endpoint(s)

I. Objective: To assess additional measure of efficacy of the regimen. To define the toxicity of the regimen in addition

II. Hypothesis: In this patient population single agent chemotherapy and pembrolizumab will provide similar efficacy but improved tolerability as 2 drug combination with pembrolizumab.

Secondary Endpoints:

I. Assess overall survival in the study population II. Assess the toxicities with the study therapy and the rate of discontinuation of study therapy due to toxicities related to study therapy

Exploratory Objective:

I. Objective: To define correlatives that can identify patients most likely to benefit from the study therapy.

II. Correlate PFS with blood-based tumor mutational burden and ctDNA.

Participants who experience confirmed disease progression or start a new anticancer therapy, will move into the Survival Follow-Up Phase and should be contacted by telephone every 12 weeks to assess for survival status until death, withdrawal of consent, or the end of the trial, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are ≥75 years of age on the day of signing informed consent with histologically confirmed diagnosis of stage IV (AJCC version 8) NSCLC with tumor PD-L1 < 50% and negative 'driver' alterations in EGFR, ALK and ROS1 will be enrolled in this study. Tumor PD-L1 expression should be assessed by FDA approved Dako 22C3 test.
2. Patients should be treatment naïve for stage IV NSCLC. Patients previously treated for earlier stages of lung cancer are eligible if they have not received systemic therapy for a minimum of 180 days prior to the start of study therapy.
3. The participant provides written informed consent for the trial.
4. Have measurable disease based on RECIST 1.1 or evaluable disease.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0,1. Evaluation of ECOG is to be performed within 7 days prior to the date of start of therapy.
6. Male participants:

   A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period.
7. Have adequate organ function as evidenced by laboratory assessment. Specimens must be collected within 10 days prior to the start of study treatment.

Exclusion Criteria:

1. Patient could not have received any anti-cancer systemic therapy for a minimum of 180 days prior to the start of study therapy. Patient should not have received prior PD-1 or PD-L1 therapy.
2. Has received prior definitive palliative radiotherapy within 2 weeks or definitive radiotherapy within 6 months of study intervention. Participants must have recovered from all radiation-related toxicities, require corticosteroids no more than 10 mg of prednisone or equivalent dose of other steroids, and not have had clinical radiation pneumonitis.
3. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
4. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
5. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
6. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. Patients with cancers such as PSA only prostate cancer may be considered after discussion with the principal investigator.

   Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ cancers
7. Has symptomatic CNS metastases and/or carcinomatous meningitis. Subjects with asymptomatic brain metastases may participate provided they are clinically stable and are not using steroids equivalent to >10mg of prednisone day prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of whether it is symptomatic or not.
8. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
10. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a known history of Human Immunodeficiency Virus (HIV) infection. Note: No HIV testing is required unless mandated by local health authority.
13. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
14. Has a known history of active TB (Bacillus Tuberculosis).
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Has had an allogenic tissue/solid organ transplant.

Ages: 75 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Median progression free survival | 6 months
  Length of time treatment to disease progression

SECONDARY OUTCOMES:
Overall survival | 12 months
  Time from progression until death

CONTACTS AND LOCATIONS:
Overall Officials: Shirish Gadgeel, MBBS, Principal Investigator — Henry Ford Health System

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will be shared with Dr. Muneesh Tewari's laboratory at University of Michigan for the CtDNA samples. Outside, of this IPD will be shared with Merck who is providing drug for this protocol. IPD will not be shared with any researchers outside of this. All subjects are assigned a study specific ID number. No direct patient identifiers leave the site.